CLINICAL TRIAL: NCT03621722
Title: AroMatherapy for Blood and Marrow Transplant PatIENTs (AMBIENT)
Acronym: AMBIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO2017-0162
Record Dates: First submitted 2018-03-21; First posted 2018-08-08 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Anxiety; Nausea; Vomiting
MeSH Terms: conditions — Anxiety Disorders; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: Patients receiving Elequil Aromatabs(treatment cohort) and patients receiving Standard of care (control cohort). In addition, patients will be receiving PRN antiemetic or PRN anxiolytics
Masking Description: The patient will be randomly assigned to a group based on their primary symptoms. The RN will be communicating with the patient for assessments, administering medications, and submitting results collected into the EPIC system.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anxiety Arm (Treatment) (Experimental): Patient will receive Elequil Aromatabs
  Interventions: Other: Elequil Aromatabs
- Nausea/Vomiting Arm (Treatment) (Experimental): Patient will receive Elequil Aromatabs
  Interventions: Other: Elequil Aromatabs
- Nausea/Vomiting Arm (Control) (No Intervention): Patient will not receive Elequil Aromatabs
- Anxiety Arm (Control) (No Intervention): Patient will not receive Elequil Aromatabs

INTERVENTIONS:
Other: Elequil Aromatabs — There will be a variety of different Aromatabs such as orange/peppermint or lavender
  Arms: Anxiety Arm (Treatment); Nausea/Vomiting Arm (Treatment)

SUMMARY:
The study is comparing the difference between the use of Elequil Aromatabs versus standard of care practice treatments on Blood Marrow Transplantation patients.

DETAILED DESCRIPTION:
The primary objective is to examine whether there are differences in the level of anxiety and nausea between patients in the treatment and control groups.

The secondary objective is to compare the number of as needed (PRN) antiemetics and anxiolytics, as well as the duration of prolonged standardized antiemetic and anxiolytic regimen for the treatment and control cohorts.

The sample size of 200 patients is anticipated to be enrolled over a period of 1 year. A total of 50 patients will be enrolled in each of the four groups The enrollment procedure will begin with a screening of patients who are admitted within 24 hours of admission for blood and marrow transplantation conditioning to evaluate if they meet the inclusion criteria. Patients who meet inclusion criteria will be offered an opportunity to participate in the study.

The patient will complete an informed consent form, then assessed to identify their predominant symptom:anxiety or nausea. Based on the patients' primary symptom, they will be randomized into either control or treatment group for a total of four groups (nausea treatment, nausea control, anxiety treatment, and anxiety control). The study will be using a Wei's Urn algorithm for the randomization sequence. The randomization sequence and patient information will be stored in a protected SharePoint folder between the 8PE and 8PW nurses enrolled with the Institutional Review Board as study staff.

Patients enrolled in the nausea control/treatment group will be required to complete a Generalized Anxiety Disorder 7-Item Scale (GAD-7) form to determine the baseline of anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Adult blood and marrow transplant patients admitted to 8 Pavilion East Blood and Marrow Transplant and 8 Pavilion West Blood and Marrow Transplant for autologous and allogeneic blood and marrow transplant conditioning (chemotherapy and/or radiation therapy) and transplant cell infusion
* Ages 22 and above. Adults ages 18-21 are admitted under the pediatric service and are not admitted to 8PE and 8PW
* Patients with blood and marrow transplant conditioning induced nausea and vomiting-
* Patients expressing feeling of anxiety
* English and Spanish speaking only
* Patients enrolled in other research studies that allow them to participate

Exclusion Criteria:

* Patients with known allergy to lavender
* Patient with known allergy to orange/peppermint
* Patients less than 22 years
* Patients with olfactory/sinus impairment
* Patients unable to give written informed consent
* Patients admitted for inpatient conditioning but receiving transplant cell infusion in the outpatient setting

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Using the Halpin 0-to-5 Nausea and Vomiting Scales to document the degree of severity of patients' self-reported blood and marrow transplant conditioning regimen induced nausea and vomiting | 12-hour intervals for a year
  Differences in the severity of nausea and vomiting between patients in the treatment and control groups
Using the Patient Self-Report of Anxiety Assessment Tool to document the degree of severity of patients' self-reported anxiety | 12-hour intervals for a year
  Differences in the severity of anxiety between patients in the treatment and control groups

SECONDARY OUTCOMES:
Number of PRN antiemetics for prolonged standardized antiemetic regimen | 1 year
  These are patients who self-report blood and marrow transplant conditioning regimen induced nausea and vomiting in the treatment and control cohorts
Duration of PRN antiemetics for prolonged standardized antiemetic regimen | 1 year
  These are patients who self-report blood and marrow transplant conditioning regimen induced nausea and vomiting in the treatment and control cohorts
Number of PRN anxiolytics for prolonged standardized anxiolytic regimen | 1 year
  These are patients who self-report blood and marrow transplant conditioning regimen induced anxiety in the treatment and control cohorts
Duration of PRN anxiolytics for prolonged standardized anxiolytic regimen | 1 year
  These are patients who self-report blood and marrow transplant conditioning regimen induced anxiety in the treatment and control cohorts
Using the Patient Self-Report of Anxiety Assessment Tool to document the severity of anxiety prior to and following application of the patch | one hour prior to and following application of the patch
  The level of anxiety in the hour prior to and following application of the patch for patients in the treatment arm
Using the Halpin 0-to-5 Nausea and Vomiting Scales to document the severity of nausea/vomiting prior to and following application of the patch | one hour prior to and following application of the patch
  The level of nausea/vomiting in the hour prior to and following application of the patch for patients in the treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Megan Tracey, MSN, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be handled in a confidential manner to meet mandated IT security standards and prevent loss of privacy. All electronic files will be stored in an encrypted and password-protected database on a secure medical center server. Any research data extracted from participants' medical records will be recorded in REDCap and electronic spreadsheets will be kept on a password protected computer. The information will be de-identified for study analysis. If the results of the trial are published, participants' identities will remain confidential and all data will be presented in the aggregate.
  Publications resulting from this research will not contain any information that could potentially identify participants, either directly or indirectly.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication